CLINICAL TRIAL: NCT07326982
Title: Efficacy of Ultrasound-Guided Interfascial Hydrodissection for Myofascial Pain Syndrome of the Gluteus Maximus in Patients With Piriformis Syndrome: A Double-Blind Randomized Controlled Trial.
Brief Title: Ultrasound-Guided Interfascial Hydrodissection for Gluteal Myofascial Pain in Piriformis Syndrome: A Prospective Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Busra Nur Aslantas, Resident Physician, Physical Medicine and Rehabilitation Department, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTFPIRHD2025
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Piriformis Syndrome; Gluteus Maximus Myofascial Pain
Keywords: Interfascial hydrodissection; Gluteal pain; Ultrasound-guided injection
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Interfascial Hydrodissection (Experimental): Ultrasound-guided interfascial hydrodissection is performed in the interfascial space between the gluteus maximus and piriformis muscles.
  Interventions: Procedure: Ultrasound-Guided Interfascial Hydrodissection
- Ultrasound-guided gluteus maximus dry needling (Active Comparator): Participants receive ultrasound-guided dry needling applied to the gluteus maximus muscle.
  Interventions: Procedure: Ultrasound-Guided Gluteus Maximus Dry Needling

INTERVENTIONS:
Procedure: Ultrasound-Guided Interfascial Hydrodissection — Ultrasound-guided interfascial hydrodissection is performed in the interfascial plane between the gluteus maximus and piriformis muscles.
  Arms: Ultrasound-Guided Interfascial Hydrodissection
Procedure: Ultrasound-Guided Gluteus Maximus Dry Needling — Ultrasound-guided dry needling is performed on the gluteus maximus muscle without fluid administration.
  Arms: Ultrasound-guided gluteus maximus dry needling

SUMMARY:
This randomized, double-blind prospective trial investigates whether ultrasound-guided interfascial hydrodissection using 10% dextrose is more effective than dry needling in treating gluteal myofascial pain coexisting with piriformis syndrome. Following diagnostic piriformis injection response, eligible patients will be randomized into two treatment arms and followed at 1 hour, 1 week, 1 month, and 3 months. The primary hypothesis is that interfascial hydrodissection will provide superior long-term analgesic outcomes due to fascial separation, neuromodulation, and nociceptor suppression.

DETAILED DESCRIPTION:
Piriformis syndrome (PS) is a neuromuscular condition characterized by compression or irritation of the sciatic nerve at the piriformis muscle level. Patients frequently present with unilateral gluteal pain that worsens with prolonged sitting, hip movement, or palpation over the piriformis locus. Although the neuropathic component of PS is attributed to sciatic nerve irritation, the somatic pain component is believed to arise from myofascial dysfunction within gluteal structures, particularly the piriformis muscle.

Recent clinical observations indicate that many patients diagnosed with PS also exhibit features of gluteus maximus myofascial pain syndrome (GM-MPS). The gluteus maximus muscle has a large fascial interface with the piriformis muscle, and nociceptive stimulation originating from this interface may contribute to persistent gluteal pain in PS. Despite this, the fascial contribution to symptom persistence remains poorly investigated, and therapeutic interventions are largely directed toward the piriformis alone.

Interfascial hydrodissection is an emerging ultrasound-guided technique in which liquid is injected between tissue planes to mechanically separate fascial layers, improve gliding, and modulate sensory nociceptive fibers. Dextrose solutions have been increasingly used in ultrasound-guided interfascial injections based on their proposed neuromodulatory and regenerative effects. However, evidence regarding its long-term efficacy in gluteal myofascial pain, particularly when coexisting with PS, is limited.

This prospective, randomized, double-blind clinical trial aims to evaluate the therapeutic effectiveness of interfascial hydrodissection using 10% dextrose solution between the gluteus maximus and piriformis muscles in patients with PS diagnosed through positive diagnostic injection response. Patients with ≥50% pain reduction one hour after diagnostic piriformis injection will be randomized into two treatment groups: (1) ultrasound-guided interfascial hydrodissection and (2) dry needling of the gluteus maximus muscle. Both interventions will be performed under ultrasound guidance to ensure accuracy and standardization.

Outcome assessment will include numerical pain scoring, percentage pain reduction, and clinical improvement at one hour, one week, one month, and three months post-intervention. The first assessor will be blinded to treatment allocation, ensuring independent measurement of outcomes. It is hypothesized that interfascial hydrodissection will provide superior long-term pain relief compared with dry needling by separating adhered fascial planes, improving local mobility, and reducing nociceptive drive through dextrose-mediated neuromodulation.

If successful, this trial will provide the first structured evidence evaluating the role of gluteus maximus-piriformis fascial interface treatment in PS and may identify an overlooked pain generator in this common syndrome. Results could expand therapeutic options for PS, support broader application of interfascial hydrodissection, and contribute to clinical understanding of fascial pain mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* Buttock pain with or without radiation to the lower extremity Positive clinical response to an ultrasound-guided diagnostic lidocaine injection of the piriformis muscle.
* Ability to understand and provide written informed consent

Exclusion Criteria:

* Active lumbar radiculopathy
* History of hip joint pathology or prior hip surgery
* Previous injection or dry needling treatment to the gluteal region within the last 3 months
* Coagulation disorders or use of anticoagulant therapy
* Pregnancy
* Local infection at the injection site
* Inability to complete the study protocol or attend follow-up visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Assessed by Numeric Rating Scale | 3 months after the intervention
  Pain intensity is assessed using the Numeric Rating Scale (NRS, 0-10) for pain at rest, during activity, at night, while standing, sitting, lying down, and for overall pain.

SECONDARY OUTCOMES:
Pain Intensity Assessed by Numeric Rating Scale | 1 week after the intervention
  Pain intensity is assessed using the Numeric Rating Scale (NRS, 0-10) for pain at rest, during activity, at night, while standing, sitting, lying down, and for overall pain.
Pain Intensity Assessed by Numeric Rating Scale | 1 month after the intervention
  Pain intensity is assessed using the Numeric Rating Scale (NRS, 0-10) for pain at rest, during activity, at night, while standing, sitting, lying down, and for overall pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data sharing has not been decided at this stage. Although ethical approval for the study has been obtained, any potential data sharing will be considered in the future upon reasonable request and in accordance with participant consent and institutional policies.

REFERENCES:
- [Result] Tantanatip A, Patisumpitawong W, Lee S. Comparison of the Effects of Physiologic Saline Interfascial and Lidocaine Trigger Point Injections in Treatment of Myofascial Pain Syndrome: A Double-Blind Randomized Controlled Trial. Arch Rehabil Res Clin Transl. 2021 Mar 9;3(2):100119. doi: 10.1016/j.arrct.2021.100119. eCollection 2021 Jun. PMID 34179755
- [Result] Misirlioglu TO, Akgun K, Palamar D, Erden MG, Erbilir T. Piriformis syndrome: comparison of the effectiveness of local anesthetic and corticosteroid injections: a double-blinded, randomized controlled study. Pain Physician. 2015 Mar-Apr;18(2):163-71. PMID 25794202
- [Result] Kaga M, Ueda T. Effectiveness of Hydro-Dissection of the Piriformis Muscle Plus Low-Dose Local Anesthetic Injection for Piriformis Syndrome: A Report of 2 Cases. Am J Case Rep. 2022 Feb 6;23:e935346. doi: 10.12659/AJCR.935346. PMID 35124689